CLINICAL TRIAL: NCT04688944
Title: The Correlation Between Degeneration of Paraspinal Muscle and Outcome of Patients With Lumbar Spinal Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019400
Record Dates: First submitted 2020-06-28; First posted 2020-12-30 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Lumbar Spinal Stenosis; Paraspinal Muscle
Keywords: degeneration of paraspinal muscle; lumbar spinal stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: (1) age ≥ 45 years, (2) diagnosed LSS through a combination of clinical history, physical examination and radiological changes showing spinal canal stenosis on magnetic resonance imaging
  Interventions: Other: observation
- healthy people: (1) age ≥ 45 years; (2) without chronic low back pain (LBP)

INTERVENTIONS:
Other: observation — observation the difference between two groups
  Groups: patients

SUMMARY:
The photographical and functional parameters of paravertebral muscle in patients with lumbar spinal stenosis will be measured to investigate the correlation between paravertebral muscle degeneration and symptoms and prognosis of patients.By measuring the parameters of paravertebral muscle with normal people, the differences between the patients and normal people will be compared to establish an appropriate paravertebral muscle evaluation method.

DETAILED DESCRIPTION:
It is a prospective observational study. This study will recruit 200 patients with lumbar spinal stenosis who will undertake posterior lumbar decompression and fusion surgery in our hospital.They all take preoperative lumbar mri examination and waist and back muscle strength test as well as recording their preoperative visual analogue scale,oswestry disability index, lumbar stiffness disability index score.All patients will receive a follow-up lasting for 1 year,and we will record patients outcomes,such as visual analogue scale,oswestry disability index and lumbar stiffness disability index score at each follow-up time. At the same time,we will recruit 100 healthy subjects without lumbar diseases or chronic lumbar pain. The difference of their age with patients was less than 5 years. Meanwhile, lumbar dorsal muscle strength test and lumbar mri examination were conducted, and visual analogue scale as well as oswestry disability index and lumbar stiffness disability index score was recorded in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* patients with lumbar spinal stenosis
* age>45 years old
* without other spinal disease
* without history of former spinal surgery

Exclusion Criteria:

* With neuromuscular diseases
* With hip joint or knee joint disease
* Acute or severe chronic back pain of spinal stenosis that could interfere with the evaluation of endurance
* Other serious diseases impacting the evaluation of endurance

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 patients with lumbar spinal stenosis and 100 healthy people
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-10-12 (Estimated); Study Completion 2024-01-21 (Estimated)

PRIMARY OUTCOMES:
cross-sectional area of paraspinal muscles | Baseline
  the cross-sectional area of paraspinal muscles reflects the quantity of paraspinal muscles. Higher cross-sectional area of paraspinal muscles means larger paraspinal muscle.
functional cross-sectional area of paraspinal muscles | Baseline
  functional cross-sectional area of paraspinal muscles reflects the quality of paraspinal muscles. It means the lean paraspinal muscle.
Performance time of paraspinal muscle endurance test | Baseine
  Participants were asked to lie prone on a plinth and lift their sternum from the plinth, raising their upper body.While maintaining this position, participants were asked to keep their arms in line with the body axis and not in contact with the plinth. Task failure was determined by a drop in the angle of trunk of greater than 10°at any point. The time was recorded until task failure or until the maximum contraction duration was reached (300 s).
lumbar stiffness disability index | the follow-up time of 3 months
  The lumbar stiffness disability index ranges from 0 to 100. Higher scores mean a worse outcome
lumbar stiffness disability index | the follow-up time of 6 months
  The lumbar stiffness disability index ranges from 0 to 100. Higher scores mean a worse outcome.
lumbar stiffness disability index | the follow-up time of 12 months
  The lumbar stiffness disability index ranges from 0 to 100. Higher scores mean a worse outcome.
lumbar stiffness disability index | Baseline
  The lumbar stiffness disability index ranges from 0 to 100. Higher scores mean a worse outcome.
The Oswestry Disability Index | Baseline
  The Oswestry Disability Index ranges from 0 to 100.Higher scores mean a worse outcome.
The Oswestry Disability Index | the follow-up time of 3 months
  The Oswestry Disability Index ranges from 0 to 100.Higher scores mean a worse outcome.
The Oswestry Disability Index | the follow-up time of 6 months
  The Oswestry Disability Index ranges from 0 to 100.Higher scores mean a worse outcome.
The Oswestry Disability Index | the follow-up time of 12 months
  The Oswestry Disability Index ranges from 0 to 100.Higher scores mean a worse outcome.
Visual Analog Score | Baseline
  Visual Analog Score is used to evaluate pain,ranging from 0 to 10.Higher scores mean a worse outcome.
Visual Analog Score | the follow-up time of 3 months
  Visual Analog Score is used to evaluate pain,ranging from 0 to 10.Higher scores mean a worse outcome.
Visual Analog Score | the follow-up time of 6 months
  Visual Analog Score is used to evaluate pain,ranging from 0 to 10.Higher scores mean a worse outcome.
Visual Analog Score | the follow-up time of 12 months
  Visual Analog Score is used to evaluate pain,ranging from 0 to 10.Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: weishi li, Study Chair — department of orthopaedic, peking university third hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided